CLINICAL TRIAL: NCT04286425
Title: Modification of Endometrial Receptivity After Vaginal Seminal Plasma Application: a Randomized Clinical Trial
Brief Title: Modification of Endometrial Receptivity After Vaginal Seminal Plasma Application
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Jens Fedder, Professor, MD, PhD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lab.Reprod.Biol. - Odense.05
Record Dates: First submitted 2020-02-14; First posted 2020-02-27 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Endometrial Receptivity
Keywords: fertility; seminal plasma; endometrium
MeSH Terms: interventions — Seeds; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 500 µl of saline solution applied in the vaginal volt twice :
  1. one month before the IVF procedure during the ovulation period
  2. Same month of the IVF procedure after ovum pick up
  Interventions: Other: saline solution
- seminal plasma (Active Comparator): 500 µl of seminal plasma applied in the vaginal volt twice :
  1. one month before the IVF procedure during the ovulation period
  2. Same month of the IVF procedure after ovum pick up
  Interventions: Other: seminal plasma

INTERVENTIONS:
Other: seminal plasma — Seminal plasma free of sperm, from donor men with normal sperm parameters, and tested for HIV1, HIV2, Hepatitis B, Hepatitis C, Syphilis, Chlamydia and Gonorrhea on blood and urine
  Arms: seminal plasma
Other: saline solution — saline solution
  Arms: Placebo

SUMMARY:
The aim of the project is to investigate the effect of seminal plasma on the endometrium and to evaluate changes in the endometrial receptivity after exposure to seminal plasma.

Implantation is still an important limiting factor for the improvement of pregnancy rate in the Assisted Reproductive Technology (ART). Usually, in fertility clinics, only the spermatozoa are used for the treatments while the rest of the seminal fluid is discarded. However, the importance of seminal fluid in fertility has gained interest in the last years but no conclusive that has been obtained yet.

Experimental group:

We decided to focus our attention on lesbian couples and single women undergoing ART procedures because they could benefice the most from this treatment since they usually do not have contact with seminal plasma. Moreover, to the best of our knowledge, they have more problems in achieving a pregnancy than heterosexual couples. Our observation is supported by a preliminary analysis of data from the Dansk fertilitetsselskab.

Design Randomized, double-blinded, placebo-controlled study

* Group 1 treated: 20 healthy lesbian or single women receiving assisted reproduction
* Group 2 control: 20 healthy lesbian or single women receiving assisted reproduction

Treatment

* One month before the IVF procedure: First seminal plasma/placebo application during ovulation period
* Same month of the IVF procedure: second seminal plasma/placebo application after ovum pick up

  5 days after the first application an endometrial biopsy and one blood sample will be taken for analysis.

Analysis:

Endometrial transcriptome microarray analysis that will be verified through protein analysis.

Differences in the transcriptome between the two groups will be compared with data in literature for an optimal endometrial receptivity. Moreover, clinical pregnancy rate and pregnancy outcome will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy lesbian and single women receiving IVF assisted reproduction treatment at OUH Fertility Clinic

Exclusion Criteria:

* Language problems to such an extent that subjects do not understand the scope of the study.
* Abnormal high follicle-stimulating hormone
* severe endometriosis,
* severe polycystic ovarian syndrome
* chronic diseases

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — It is a study on endometrial factors in female infertility
Enrollment: 40 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Endometrial transcriptome profile: mRNA array (fold change) | 24 months
  mRNA array ( fold change). Endometrial mRNA expression will be compared between treated and control group mRNA expression expression will be compared between treated and control group mRNA expression profiles will be compared with literature data for an optimal endometrial receptivity.
Endometrial protein concentration of leukemia inhibitory factor (LIF) | 24 months
  LIF concentration measured by ELISA test. LIF concentration will be compared between treated and control group. LIF has been chosen for its importance in implantation.

SECONDARY OUTCOMES:
Endometrial proteins concentration | 24 months
  protein concentration of relevant genes selected after transcriptome analysis will be measured using ELISA test. Proteins concentration will be compared between treated and control group.
clinical pregnancy rate | 6 months
  clinical pregnancy rate difference between treated and control group ( presence of a fetal heartbeat at 6-7 weeks of pregnancy)
pregnancy rate | 12 months
  pregnancy rate difference between treated and control group (number of live birth)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Andrology & Fertility Clinic, Department D, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No